CLINICAL TRIAL: NCT04999579
Title: Digital Occlusal Analysis of Ultra Suction Retained Complete Denture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Shady El Naggar, Dr, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 1122110085
Record Dates: First submitted 2020-12-31; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Complete Edentulism

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complete denture (Active Comparator): Conventional complete denture without supporting devices
  Interventions: Device: T scan
- Ultra suction retained complete denture (Experimental): Conventional complete denture with ultra suction device
  Interventions: Device: T scan

INTERVENTIONS:
Device: T scan — Occlusal load analysis

SUMMARY:
Bite testing using T-Scan allows the evaluation of occlusal contacts prior to making a bite adjustment. The T-Scan can indicate premature contact and the load distribution on teeth, and provide measurable force and time information that ensures proper occlusal adjustment.

DETAILED DESCRIPTION:
Prior to employing T-Scan occlusal analyzer to assess the occlusion on the complete denture, complete denture was seated and checked for fitness, stability, pressure areas with pressure indicating paste and border evaluation and extension. The peripheral seal should be evident so that the denture-maintained suction against maxillary tissues. Upon completion of these fit and stability assessments, the occlusion could then be addressed.

The method considered for the occlusal analysis was a computerized system . The system was composed of a computer with a specific board and software capable of converting information recorded by the sensor to visual and numerical information on tooth contact. For Tekscan system to function properly, computer system must meet or exceed specified system requirements.

The Tekscan USB handle, does not require an additional interface card or parallel box in order tobe connected to computer. When inserted into computer, the computer's operating system will automatically detect and configure the hardware for use. The T-Scan sensor was an ultra-thin (.004", 0.1 mm), flexible printed circuit that detected the patient's occlusal parameters.

ELIGIBILITY:
Inclusion Criteria:

* All implant indicated.

Exclusion Criteria:

* All implant contraindicated

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Occlusal load analysis | One year
  occlusal load analysis of the ultra suction system in complete denture being evaluated by T-scan system

CONTACTS AND LOCATIONS:
Overall Officials: El Naagar, Principal Investigator — Badr university in Cairo
Locations (1):
- Badr university in Cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-08-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT04999579/Prot_SAP_ICF_000.pdf